CLINICAL TRIAL: NCT00665873
Title: Antibiotic Therapy is Not Necessary to Implant Totally Implantable Venous Access Devices: Randomized Prospective Study
Acronym: TIVAD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universita degli Studi di Catania (Other)
Responsible Party: Isidoro DI CARLO, MD, PhD, FACS, University of Catania
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1-28064152
Record Dates: First submitted 2008-04-02; First posted 2008-04-24 (Estimated); Last update posted 2008-05-08 (Estimated); Status verified 2008-05

CONDITIONS: Infections
Keywords: Totally Implantable Venous Access Devices; Infections; Chemotherapy; Valuated infections TIVAD
MeSH Terms: conditions — Infections | interventions — Vascular Access Devices; Amoxicillin-Potassium Clavulanate Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): Antibiotics
  Interventions: Device: PORT-A-CATH (Smiths Medical Inc., MN); Drug: Amoxicillin and clavulanic acid
- B (Active Comparator): No Antibiotics
  Interventions: Device: PORT-A-CATH (Smiths Medical Inc., MN)

INTERVENTIONS:
Device: PORT-A-CATH (Smiths Medical Inc., MN) — Port a Cath implanted by surgical cut-down
  Other Names: Totally implantable venous access device (TIVAD)
Drug: Amoxicillin and clavulanic acid — 1 gr i.v. before the procedure
  Other Names: Antibiotics vs no antibiotics
  Arms: A

SUMMARY:
BACKGROUND: The growing use of totally implantable venous access devices (TIVAD) has caused the simultaneous increase of various complications. The infection of the TIVAD or the subcutaneous pocket in which the device is positioned is one of the most encountered complications. The aim of this study is to evaluate the role of the antibiotic in the prevention of the infection of the surgical site and the TIVAD until 30 days after the implant.

METHODS: The authors enrolled one hundred consecutive patients divided into two randomized arms: group A (antibiotic), group B (no antibiotic), each of 50 patients. All the patients were affected by solid tumors needing chemotherapy continuously. TIVADs were implanted surgically in cephalic vein. Signs or symptoms considered were: pain, localized swelling, redness, and heat. White cell count was considered on the first, third, and seventh postoperative days, and the tests were made in the in-hospital laboratory. Body temperatures were checked twice daily for 7 days.

DETAILED DESCRIPTION:
PATIENTS AND METHODS One hundred consecutive patients were enrolled for the present study from January 2004 to September 2006. The patients were divided into two arms, each of 50 patients, and they were randomized using sealed envelopes that were opened only in the operating room 30 min before the start of the procedure. All the patients were aged more than 18 years and were affected by solid tumors. In all the patients, the TIVAD was necessary to infuse chemotherapy continuously. The type of device utilized in all patients was composed of a catheter of polyurethane and a titanium portal reservoir covered with polysulfone (PORT-A-CATH, Smiths Medical Inc., MN).

Age, gender, comorbidity (cardiovascular, pulmonary, renal, hepatic, coagulopathy, diabetes), white cells, platelets, prothrombin time (less than 70%), kind of tumoral disease, numbers of chemotherapeutical cures before the surgical procedure, experience of surgeons (resident or surgeon), preparation of the skin of the patients, time and kind of hand scrub of the surgeons, kind of antibiotic used, and time of administration were considered for the present study. All the devices were implanted in the operating room using the cephalic vein dissected surgically; the technique used has been previously described.3 White cell count was considered on the first, third, and seventh postoperative days, and the tests were made in the in-hospital laboratory. Body temperatures were checked twice daily for 7 days. Eight days after the surgical procedure, sutures of the skin were removed. The skin wound was covered with a sterile drape until the ninth postoperative day. After this time, the patients used any skin protection, but the skin wound was checked one time each week for a total of 30 days. All the devices were used to infuse chemotherapy drugs 10 days after the surgical procedure. From the 10th to the 30th days, the devices were used, at minimum, one time.

A single dose of cephalosporin (1 gr of amoxicillin and clavulanic acid ) was administered intravenously 10 min before the skin incision.

For the surgical site infections (SSI), the criteria of the Centers for Disease Control and Prevention (CDC), Atlanta, Georgia,9 were applied. By these criteria, SSIs are classified as being either incisional or organ/space. Incisional SSIs are further divided into those involving only skin and subcutaneous tissue (superficial incisional SSI) and those involving deeper soft tissues of the incision (deep incisional SSI). Organ/space SSIs involve any part of the anatomy (e.g., organ or space) other than incised body wall layers that was opened or manipulated during the operation (Fig. 1).

The following signs or symptoms for defining a superficial incisional infection were considered: pain, localized swelling, redness, and heat.9 Infection was considered if these signs and symptoms occurred within 30 days after the surgical procedure, and the end points were considered to be a body temperature more than 37.5°C, white cells more than 11,000 K/æL, and one or more of the following signs: pain, localized swelling, redness, or heat.

The state of the skin was evaluated in people with the same surgical team, which was composed of the surgeons (one skilled, with more than 400 previous procedures, and one resident, with 20 previous procedures) and two nurses.

Following these rules, depending on the results of a computer-generated randomization enclosed in sealed envelopes, 100 patients were divided into two groups of 50 patients: group A (patients were submitted to the short-term prophylaxis with cefalosporin 10 min before skin incision) and group B (patients without any antibiotic prophylaxis). All the patients were hospitalized the night after the surgical procedure. A statistical study, to compare the means and standard deviations of each group, was performed using Student's t-test (independent, two-sided).

ELIGIBILITY:
Inclusion Criteria:

* Age
* Gender
* Comorbidity
* White cells
* Platelets
* Prothrombin time
* Any kind of tumoral disease
* Numbers of chemotherapeutical cures before the surgical procedure
* Experience of surgeons
* Preparation of the skin of the patients
* Time and kind of hand scrub of the surgeons
* Kind of antibiotic used, and time of administration.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2004-01; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)